CLINICAL TRIAL: NCT04736927
Title: An Open-label, Fixed-sequence, Drug-drug Interaction Study in Healthy Subjects to Evaluate the Effect of GLPG3667 on the Pharmacokinetics of Midazolam, a Sensitive Index Substrate of CYP3A4
Brief Title: Drug-drug Interaction Study With GLPG3667 and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-105; 2020-004846-12 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLPG3667 + Midazolam (Experimental)
  Interventions: Drug: GLPG3667; Drug: Midazolam

INTERVENTIONS:
Drug: GLPG3667 — From Day 3 to Day 8, GLPG3667 capsules q.d. orally in fed state.
Drug: Midazolam — On Day 1 and Day 7 as liquid formulation, orally in fed state.

SUMMARY:
A study in healthy volunteers to look at the effect of the test medicine, GLPG3667, on how midazolam (MDZ) is taken up and eliminated by the body.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (extremes included), on the date of signing the informed consent form. Female subjects should be of non-childbearing potential, defined as permanently surgically sterile (bilateral oophorectomy, i.e. surgical removal of ovaries, bilateral salpingectomy, i.e. surgical removal of the fallopian tubes, or hysterectomy, i.e. surgical removal of uterus), or with no menses for 12 or more months without an alternative medical cause AND a follicle-stimulating hormone level in the postmenopausal range. These female subjects must also have a negative pregnancy test. For surgical sterilization, documented confirmation will be requested.
* A body mass index between 18.0 and 30.0 kg/m², inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests available at screening and prior to enrolment. Neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Total bilirubin, aspartate aminotransferase, and alanine aminotransferase must be within normal ranges. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to investigational product (IP) and/or MDZ ingredients or history of a significant allergic reaction to IP and/or MDZ ingredients as determined by the investigator.
* Treatment with any medication (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy for postmenopausal subjects) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of MDZ | From Day 1 until Day 9
  To determine the effect of GLPG3667 on the pharmacokinetics (PK) of MDZ.
Maximum observed plasma concentration (Cmax) of MDZ | From Day 1 until Day 9
  To determine the effect of GLPG3667 on the PK of MDZ.

SECONDARY OUTCOMES:
Cmax of GLPG3667 | From Day 3 until Day 8
  To evaluate the PK of GLPG3667 in the presence of a single dose of MDZ.
Area under the plasma concentration-time curve over the dosing interval (AUCτ) for GLPG3667 | From Day 3 until Day 8
  To evaluate the PK of GLPG3667 in the presence of a single dose of MDZ.
Trough plasma concentration observed (Ct) for GLPG3667 | From Day 3 until Day 8
  To evaluate the PK of GLPG3667 in the presence of a single dose of MDZ.
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From Day 1 through study completion, an average of 3 weeks
  To evaluate the safety and tolerability of GLPG3667 alone or when coadministered with MDZ.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rueda-Rincon, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No